CLINICAL TRIAL: NCT03882918
Title: An Open-Label Study to Evaluate the Long-Term Safety, Tolerability, and Efficacy of OV101 in Individuals With Angelman Syndrome
Acronym: ELARA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision
Sponsor: Healx AI (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OV101-18-002
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Angelman Syndrome
MeSH Terms: conditions — Angelman Syndrome | interventions — gaboxadol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OV101 (Experimental): once daily at bedtime (gaboxadol)
  Interventions: Drug: OV101

INTERVENTIONS:
Drug: OV101 — Each subject will be titrated to his or her maximal tolerated daily dose, up to a maximum daily dose of 15 mg at bedtime.
  Other Names: gaboxadol

SUMMARY:
This open-label study (OV101-18-002) will evaluate the long-term (52 weeks) safety of OV101 in subjects with AS and provide additional OV101 treatment to those subjects who completed Study OV101-15-001 (NCT02996305). Subjects with AS who completed the pharmacokinetic Study OV101-16-001 (NCT03109756) will also be permitted to participate, provided they meet all entry criteria.

DETAILED DESCRIPTION:
This will be an open-label, long-term safety study for evaluation of further treatment with OV101 in subjects with AS who have completed previous Ovid studies (OV101-15-001 or OV101-16-001). There will be no placebo treatment. As this study will enroll subjects who have completed previous AS studies for different periods of time before entering this study, subjects will be required to complete screening and baseline visits before receiving OV101 under this protocol.The secondary objective of this study is to evaluate the long-term efficacy of OV101 treatment assessed by changes in behavior, sleep, and functioning in individuals with AS.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all the following criteria to be enrolled in this study:

1. Has completed the OV101-15-001 or OV101-16-001 study up to the EOS.
2. Is male or female and 13 to 49 years old (inclusive) at the time of inclusion in the OV101-15-001 or OV101-16-001 study.
3. Has a previous diagnosis of AS with molecular confirmation from the OV101-15-001 or OV101-16-001 study.
4. Has an LAR/caregiver capable of providing informed consent and able to attend all scheduled study visits, oversee the administration of study drug, and provide feedback regarding the subject's symptoms and performance as described in the protocol.
5. Provides assent to the protocol (to the extent possible and in accordance with local institutional review board (IRB) and regulatory requirements) and has an LAR/caregiver who will provide written informed consent. Subjects providing assent must do so at the same visit as LAR/caregiver written informed consent is provided.
6. Can swallow study drug capsules or ingest the contents of study drug capsules after sprinkling the capsule contents onto 1 spoon of applesauce or low-fat yogurt.
7. Is currently receiving a stable dose of concomitant medications such as anti-epileptic medication, gabapentin, clonidine, trazadone, melatonin, and special diets for at least 4 weeks prior to Baseline.
8. Agrees to remain sexually abstinent from the first day of screening until 30 days after the last dose of study treatment.
9. Has LAR/caregiver(s) who agree not to post any of the subject's personal medical data or information related to the study on any website or social media site (eg, Facebook, Instagram, Twitter) until notified that the study is completed.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Discontinued from the OV101-15-001 or OV101-16-001 study due to safety reasons causally related to OV101.
2. Has a concomitant disease (eg, gastrointestinal, renal, hepatic, endocrine, respiratory, or cardiovascular system disease) or condition or any clinically significant finding at Screening that could interfere with the conduct of the study or that would pose an unacceptable risk to the subject in this study.
3. Has poorly controlled seizures defined as > 3 seizures lasting < 3 minutes per week or > 1 seizure episode lasting more than 3 minutes per week or as per medical monitor judgment.
4. Has clinically significant clinical laboratory abnormalities or vital signs at the time of screening (eg, alanine aminotransferase or aspartate aminotransferase > 2.5 × upper limit of normal; total bilirubin or creatinine > 1.5 × upper limit of normal). Retesting of clinical laboratory parameters may be allowed after consultation with the medical monitor or designee.
5. Current use of benzodiazepines, zolpidem, zaleplon, zopiclone, eszopiclone, barbiturates, or ramelteon for sleep within the 4 weeks prior to Day 1. Benzodiazepines administered for situational anxiety related to occasional procedures or events are permitted.
6. Has a history of suicidal behavior or is considered by the investigator to be at increased risk of suicide.
7. Has any condition or circumstance that, in the opinion of the investigator, makes the subject unsuitable for enrollment.
8. Has enrolled in any clinical trial or used any investigational agent or device, or has participated in any investigational procedure, within the 30 days before screening or does so concurrently with this study.
9. Is a family member of the investigator or of study site staff.

Ages: 13 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 141 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (10):
  - Ovid Therapeutics Investigative Site, Phoenix, Arizona
  - Ovid Therapeutics Investigative Site, San Diego, California
  - Ovid Therapeutics Investigative Site, Atlanta, Georgia
  - Ovid Therapeutics Investigative Site, Chicago, Illinois
  - Ovid Therapeutics Investigative Site, Boston, Massachusetts
  - Ovid Therapeutics Investigative Site, Lexington, Massachusetts
  - Ovid Therapeutics Investigative Site, Cincinnati, Ohio
  - Ovid Therapeutics Investigative Site, Media, Pennsylvania
  - Ovid Therapeutics Investigative Site, Nashville, Tennessee
  - Ovid Therapeutics Investigative Site, Tacoma, Washington
- Ovid Therapeutics Investigative Site, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heussler HS. Emerging Therapies and challenges for individuals with Angelman syndrome. Curr Opin Psychiatry. 2021 Mar 1;34(2):123-128. doi: 10.1097/YCO.0000000000000674. PMID 33395098

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OV101
Started | 141
Completed | 1
Not Completed | 140
Not completed — Study terminated by sponsor | 98
Not completed — Protocol Violation | 1
Not completed — Other | 9
Not completed — Lack of Efficacy | 14
Not completed — Adverse Event | 13
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: Only 1 patient completed the study, and the study was terminated early.
Arm/Group | OV101
Number analyzed (Participants) | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 100
  Between 18 and 65 years | 41
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 5
  White | 127
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 103
  Israel | 19
  Netherlands | 4
  Germany | 6
  Australia | 9

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Participants Experiencing Adverse Events in Active Treatment Group
Description: Safety assessments related to the primary study objective of evaluating the safety and tolerability of OV101, including serious adverse events (SAEs) and adverse events (AEs) leading to study discontinuation, as assessed by the number of participants who experienced at least one adverse event.
Time Frame: Change from baseline to Week 39
Population: One participant completed the study; all other participants did not complete the study due to the early termination of the study by the Sponsor.
Measure: Number; unit: participants
Arm/Group | OV101
Number analyzed (Participants) | 1
participants | 1

2. Secondary Outcome: To Evaluate the Long-term Efficacy of OV101 Treatment as Assessed by Changes in Behavior in Study Participants With AS Who Were at Least 4 Years Old.
Description: The long-term efficacy of OV101 was assessed by changes in irritability using the Aberrant Behavior Checklist - Irritability subscale (ABC-I), part of the broader ABC-Community (ABC-C). The final value reflects change from baseline to early termination at 39 weeks. The ABC-I consists of 15 items measuring behaviors such as aggression, self-injury, temper tantrums, and mood instability. Each item is rated by a caregiver on a 4-point scale: 0 = not at all a problem; 1 = slight problem; 2 = moderately serious; 3 = severe. Scores range from 0 (no symptoms) to 45 (maximum severity). A higher total score indicates greater behavioral disturbance and worse clinical status. The scale provides a standardized means to track symptom changes over time, making it suitable for evaluating treatment efficacy in neurodevelopmental and neuropsychiatric disorders.
Time Frame: change from baseline to 12 wks and baseline to early termination of the study at 39 weeks
Population: 132 participants were evaluated using the ABC-I.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OV101
Number analyzed (Participants) | 132
score on a scale
  Week 12 | -0.7 (1.5)
  Week 39: number analyzed (Participants) | 50
  Week 39 | -0.5 (1.3)

ADVERSE EVENTS:
Time Frame: from baseline to Week 39, as the trial was terminated early
Arm/Group | OV101
All-Cause Mortality (participants affected / at risk) | 0/141
Serious Adverse Events (participants affected / at risk) | 18/141
Other Adverse Events (participants affected / at risk) | 0/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OV101 (N=141)
Cardiac arrest (Cardiac disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Hematemesis (Gastrointestinal disorders) | 1 (1)
Corona virus infection (Infections and infestations) | 2 (2)
Device related infection (Infections and infestations) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Dehydration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Partial Seizures (Nervous system disorders) | 2 (2)
Generalized tonic-clonic seizure (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Seizure Cluster (Nervous system disorders) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Atelectasis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT03882918/Prot_SAP_001.pdf